CLINICAL TRIAL: NCT06286410
Title: Accommodation Response in Hypermetropic Anisometropia (ARIHA) Study: Accommodation Changes During Amblyopia Treatment and Pilot Residual Amblyopia Treatment Study
Brief Title: Accommodation Response in Hypermetropic Anisometropia (ARIHA Study)
Acronym: ARIHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 184950
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-02

CONDITIONS: Anisometropic Amblyopia; Accommodation Disorder
Keywords: Anisometropia; Amblyopia; Anisometropic Amblyopia; Accommodation; Plusoptix PowerRefractor 3; Anti-accommodation; Anisometropic accommodation
MeSH Terms: conditions — Amblyopia; Anisometropia

STUDY DESIGN:
Intervention Model Description: During Phase 2 of the study:
  The participants found to have residual amblyopia following standard care treatment (completed treatment but still have unequal vision) and asymmetrical accommodation (following their PR3 measurements and data interpretation), will be offered an intervention dependent upon their type of asymmetrical accommodation. There will not be any cross over in the treatment arms, and no randomisation during this pilot study, as the interventions differ and are bespoke to each patient.
  Asymmetrical accommodation can be one of two things: Aniso-A and Anti-A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aniso-A (Experimental): Aniso-A
  Those found to have anisometropic accommodation response do not focus effectively in their amblyopic eye when looking at the 0.33m (near) targets. Aniso-A response will be determined by their interocular difference in measurements at near (0.33m).
  They will be given a prescription for D-28 segment bifocal glasses. The distance section of the glasses will match their current glasses, and the bifocal add will be equivalent to the mean amount they are under accommodating by at 0.33m in their amblyopic eye during the cue conditions with glasses. Bifocals will only be worn during patching. They will wear their own current glasses for all other times. This will be made very clear to parents/caregivers, and written instructions will be given.
  The participant will act as their own controls: visual acuity at recruitment will be used to compare to visual acuity during and after the intervention.
  Interventions: Other: Bespoke glasses prescription worn during amblyopia treatment.
- Anti-A (Experimental): Anti-A
  Those found to have anti-accommodation over-accommodate in their amblyopic eye for the 2m (distance) target. Aniso-A response will be determined by their interocular difference in measurement in the distance (2m).
  They will be given a prescription for single vision distance glasses. The distance prescription in their non-amblyopic eye will be the same as their current glasses. The distance prescription in their amblyopic eye will be reduced by the same amount they are over-accommodating by during the cue conditions with glasses. This amended distance prescription will only be worn during patching. They will wear their own current glasses for all other times. This will be made very clear to parents/caregivers, and written instructions will be given.
  The participant will act as their own controls: visual acuity at recruitment will be used to compare to visual acuity during and after the intervention.
  Interventions: Other: Bespoke glasses prescription worn during amblyopia treatment.

INTERVENTIONS:
Other: Bespoke glasses prescription worn during amblyopia treatment. — The investigators aim to use the information they gather about a participant's accommodation response to be used in a bespoke glasses prescription that will be worn during amblyopia treatment. This is to try and improve vision in those with residual amblyopia following standard amblyopia treatment.

SUMMARY:
Anisometropic amblyopia is when one eye has a much stronger glasses prescription than the other, causing poor vision in one eye, even with glasses, because the brain favours the better-seeing eye.

With standard care treatment (glasses plus either patching or atropine drops given to the better seeing eye), 35% of children with anisometropic amblyopia do not have any significant visual improvements, and will have reduced vision in one eye for life. There is no consensus for the reasons why some children do not respond as well as others.

Recent research using the Plusoptix PowerRefractor (PR3), which quickly measures eye focusing (accommodation), suggested that in children with anisometropic amblyopia, the focusing of the amblyopic eye might influence treatment success. However, such measurements weren't previously common due to equipment limitations in clinics.

The investigators aim to use the non-invasive PR3 to assess accommodation in hypermetropic anisometropic amblyopia, at the University of Sheffield. This will be a two-phase study of children aged 4-10 years who have hypermetropic anisometropia. The investigators will recruit participants attending the Ophthalmology Department at Sheffield Children's NHS Foundation Trust (SCH). The investigators will take repeated measurements of accommodation at points during standard care treatment (phase 1) and conduct a pilot intervention study (phase 2) to determine whether adjusting glasses prescriptions based on accommodation responses with amblyopia treatment can improve vision in the weaker eye. The goal is to gather evidence to inform a future larger multicentre RCT to improve the visual outcomes for anisometropic amblyopic children in the future.

DETAILED DESCRIPTION:
This is a two-phase study of children aged 4-10 years who have hypermetropic anisometropia:

1. Phase 1 is a cohort observational study. It will involve repeated measurements of accommodation response (using the PR3) of hypermetropic anisometropic children during their standard care treatment at SCH. PR3 measurements (all non-invasive) will be taken at various stages of their treatment to track if accommodation responses change over time.
2. Phase 2 is a pilot intervention study. It will recruit hypermetropic anisometropic children who have finished their standard care treatment at SCH but have not achieved equal (or nearly equal) vision for initial screening. Those who are found to have asymmetrical accommodation responses, and also have residual amblyopia (unequal vision in the two eyes) will be invited to the intervention study. Bespoke glasses will be issued, based on accommodation response, and children will restart occlusion (patching) for 12 weeks while wearing the bespoke glasses. This is to assess whether a glasses adaptation based on accommodation response will help to further improve vision in their amblyopic eye.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* 4-10 years (at recruitment)
* Have hypermetropic anisometropia with ≥1.00D of difference (in spherical equivalent)
* Are currently undergoing treatment for hypermetropic anisometropia (including refractive adaptation and/or occlusion treatment - patching or atropine)
* Visual acuity in non-amblyopic eye ≤0.200 logMAR
* Any level of VA in amblyopic eye (worse than non-amblyopic eye)
* No manifest strabismus
* Accept microT with/without identity
* No other eye conditions as cause of amblyopia (e.g. stimulus deprivation amblyopia/strabismic amblyopia)
* No significant health conditions that would impact vision or accommodation response (e.g. Down's Syndrome/Cerebral Palsy)
* Informed consent from parent / guardian and assent from child (over 5 years)

Phase 2

* 4-10 years (at recruitment)
* Hypermetropic anisometropic amblyopes ≥1.00D of difference (in spherical equivalent)
* Finished standard amblyopia occlusion treatment (including patching and/or atropine)
* Asymmetric accommodation responses (Anti-A and Aniso-A) following preliminary assessment
* VA in non-amblyopic eye ≤0.200 logMAR
* Residual amblyopia (defined as interocular difference of ≥0.2 log units)
* No manifest strabismus
* Accept microT with/without identity
* No other eye conditions as cause of amblyopia (e.g. stimulus deprivation amblyopia/strabismic amblyopia)
* No significant health conditions that would impact vision or accommodation response (e.g. Down's Syndrome/Cerebral Palsy)
* Informed consent from parent / guardian and assent from child (over 5 years)

Exclusion Criteria:

Phase 1 and Phase 2

* Not within the age range 4-10 years at time of recruitment
* Has myopic anisometropia (either eye)
* <1.00D of hypermetropic anisometropia
* Vision in non-amblyopic eye worse than >0.200 logMAR
* Has a manifest strabismus
* Has amblyopia caused by an eye condition (e.g. stimulus deprivation amblyopia/strabismic amblyopia)
* Has a significant health condition that would impact vision or accommodation response (e.g. Down's Syndrome/Cerebral Palsy)
* Parent /guardian unable to give informed consent
* Parent/guardian unable to communicate in English sufficiently to give informed consent
* (Phase 2 only) does not have residual amblyopia (has equal vision in both eyes)
* (Phase 2 only) has symmetrical accommodation on the PR3 tests

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity | 12 weeks
  The change found in level of visual acuity pre- and post- pilot intervention in the amblyopic eye (phase 2).

SECONDARY OUTCOMES:
Change in PR3 accommodation measurements | 12 weeks
  The changes in PR3 accommodation measurements during standard care treatment in hypermetropic anisometropic amblyopia and the amount of participants found to have asymmetrical accommodation and residual amblyopia (both Phase 1).

CONTACTS AND LOCATIONS:
Overall Officials: Holly Geraghty, Principal Investigator — University of Sheffield
Locations (1):
- Division of Ophthalmology & Orthoptics, School of Allied Health Professions, Nursing and Midwifery, The University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No